CLINICAL TRIAL: NCT06669858
Title: Effect of Osteopathy Medicine on Post-surgical Management of Lumbosacral Arthrodesis, a Pilot Study
Brief Title: Effect of Osteopathy Medicine on Post-surgical Management of Lumbosacral Arthrodesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Européen d'Enseignement Supérieur de l'Ostéopathie de Lyon (Other)
Collaborators: Institut de la Colonne Vertébrale Lyon Charcot (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/0219L10/0219L17
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Arthrodesis; Post-operative Care; Manual Therapy; Lumbar Spine Surgery
MeSH Terms: conditions — Ankylosis | interventions — Musculoskeletal Manipulations; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual therapy standardized protocol group (Experimental): This arm received 2 session of manual therapy (standardized protocol) 2-4 days after surgery and 90 days after surgery
  Interventions: Other: manual therapy
- Sham protocol group (Sham Comparator): The sham group received a standardized protocol of ligth touch with wide pressure of the 2 hands, without intention to treat.
  Interventions: Other: Sham

INTERVENTIONS:
Other: manual therapy — In first session 6 techniques were applied to favorise fluids circulation, respiratory mecanism end equilibration of pressions (all were external soft tissue techniques, without manipulation): on cervico dorsal hinge, on cranial diaphragm, on thoracic diaphragm, on pelvic diaphram, on liver and spleen organ, on lumbar fasciae.
  In second session 6 techniques were applied in order to improve quality and quantity of legs and pelvis mobility (all were external sof tissue techniques, without manipulation) : on cervico dorsal hinge, on cranial diaphragm, on thoracic diaphragm, on pelvic diaphram, on pubic symphysis, on legs and pelvis and on lumbar fasciae
  Arms: Manual therapy standardized protocol group
Other: Sham — Wide ligth touch pressure applied with the 2 hand at day 2-4 and day 90
  Arms: Sham protocol group

SUMMARY:
Introduction : Low back pain represents a major public health issue. In some cases, surgery may be necessary, but it is not without consequences. Among these, we find pain that may require management in specialized centers as well as functional disability, particularly in cases of arthrodesis, thereby affecting the quality of life of patients. Objectives : To study the effectiveness of osteopathy in the post-surgical management of lumbo-sacral arthrodesis. Methods : A pilot study including 35 patients who underwent lumbo-sacral arthrodesis divided into 2 groups: standardized osteopathic treatment and sham. The protocol consists of 2 post-operative sessions (D2 3 and D90). The evaluated criteria were pain intensity using the VAS, functional disability with the Oswestry questionnaire, anxiety and depression with the HAD questionnaire, and analgesic consumption. Result : Compared to the sham group, the osteopathic treatment group exhibited a lack of significance in the VAS (p= NS), Oswestry (p= NS) and HAD (p= NS) scores. Analgesic consumption also demonstrated a lack of statistical significance (p= NS). Discussion : In this study, osteopathy did not show an impact on HAD, Oswestry, VAS scores, or analgesic consumption. Based on other articles, there seems to be a link between the effectiveness of osteopathy and the frequency of sessions. Thus, it might be interesting to repeat the study with a larger sample size, the use of other measurement tools, and an increase in session frequency to validate these results.

ELIGIBILITY:
Inclusion Criteria:

* having surgery in Institut de la Colonne Vertébrale
* surgery of lumbosacral arthrodesis

Exclusion Criteria:

* spine deformation
* inflammatory rhumatim
* neurodegenerative pathology
* cognitive trouble
* neoplasic pathology
* surgery complication
* second surgery
* out of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Analogic Visual Scale of pain | at day 0 pre surgery, day 2 post surgery, day 90 post surgery (pre and post intervention) and day 105 post surgery
  Pain scale from 0 (no pain) to 10 (maximal pain).

SECONDARY OUTCOMES:
OSWESTRY | day 0 pre surgery - day 90 post surgery - day 105 post surgery
  quality of life questionnary to evaluate fonctional incapacity. Score from 0 (no invalidity) to 50 (complete invalidity)
Hospital Anxiety and Depression | day 0 pre surgery, day 90 post surgery
  questionnary about depression and anxiety during hospitalisation. Score from 0 (no trouble) to 21 (severe trouble)
Antalgic consumption | from day 0 to day 105
  week table of antalgic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Laurianne Tournier-Pinloche, PhD, MsC, Osteopathe DO, Study Director — Centre Européen d'Enseignement Supérieur de l'Ostéopathie de Lyon; Pierre Grobost, PhD, Study Chair — Institut de la Colonne Vertébrale Lyon Charcot; Aline Rollet, Ostéopathe DO, MsC Cand., Principal Investigator — Centre Européen d'Enseignement Supérieur de l'Ostéopathie de Lyon
Locations (1):
- Institut de la Colonne Vertébrale Lyon Charcot, Ste Foy Les Lyons, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: beginning 3 months and ending 3 years after publication of results
Access Criteria: on demand near to the principal investigator